CLINICAL TRIAL: NCT02984956
Title: Hypotension Relationship With Pleth Variability Index In Hip Fracture Patients Who Underwent Spinal Anesthesia
Brief Title: Pleth Variability Index and Hypotension
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: ERZINCAN UNIVERSITY 4
Record Dates: First submitted 2016-12-04; First posted 2016-12-07 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Hypotension; Pleth Variability Index
Keywords: Hypotension; Pleth variability index; Hip Fracture; Spinal anesthesia
MeSH Terms: conditions — Hypotension; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: pleth variability index

SUMMARY:
Correct assessment of a patient's volume status is the most important goal for an anesthetist. However, most of the variables used for fluid response evaluation are invasive and technically challenging.Pulse oximeter is a non-invasive, standardized and widely used monitoring method in many countries. Our aim in this study is to investigate the usefulness of the noninvasive pleth variability index to predict hypotension in orthopedic hip fracture patients who underwent spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* over 65 years old
* Patients to undergo spinal anesthesia

Exclusion Criteria:

* Patients under 65 years old
* Patients to undergo general anesthesia or only sedation
* Patients with cardiac arrhythmia
* Patients with low ventricular ejection fraction
* Heart valve disease patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who underwent spinal anesthesia for hip fracture
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Detecting pleth variability index-hypotension relationship | one year

SECONDARY OUTCOMES:
pleth variability index response to fluid management | one year
Make a differential diagnosis of hypotension with pleth variability index | one year
Correlation between arterial hemoglobin and pleth variability index hemoglobin | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar A, Anel R, Bunnell E, Habet K, Zanotti S, Marshall S, Neumann A, Ali A, Cheang M, Kavinsky C, Parrillo JE. Pulmonary artery occlusion pressure and central venous pressure fail to predict ventricular filling volume, cardiac performance, or the response to volume infusion in normal subjects. Crit Care Med. 2004 Mar;32(3):691-9. doi: 10.1097/01.ccm.0000114996.68110.c9. PMID 15090949
- [Background] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Background] Preisman S, Kogan S, Berkenstadt H, Perel A. Predicting fluid responsiveness in patients undergoing cardiac surgery: functional haemodynamic parameters including the Respiratory Systolic Variation Test and static preload indicators. Br J Anaesth. 2005 Dec;95(6):746-55. doi: 10.1093/bja/aei262. PMID 16286349
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Derichard A, Robin E, Tavernier B, Costecalde M, Fleyfel M, Onimus J, Lebuffe G, Chambon JP, Vallet B. Automated pulse pressure and stroke volume variations from radial artery: evaluation during major abdominal surgery. Br J Anaesth. 2009 Nov;103(5):678-84. doi: 10.1093/bja/aep267. Epub 2009 Sep 29. PMID 19797246
- [Background] Solus-Biguenet H, Fleyfel M, Tavernier B, Kipnis E, Onimus J, Robin E, Lebuffe G, Decoene C, Pruvot FR, Vallet B. Non-invasive prediction of fluid responsiveness during major hepatic surgery. Br J Anaesth. 2006 Dec;97(6):808-16. doi: 10.1093/bja/ael250. Epub 2006 Sep 16. PMID 16980709
- [Background] Cannesson M, Delannoy B, Morand A, Rosamel P, Attof Y, Bastien O, Lehot JJ. Does the Pleth variability index indicate the respiratory-induced variation in the plethysmogram and arterial pressure waveforms? Anesth Analg. 2008 Apr;106(4):1189-94, table of contents. doi: 10.1213/ane.0b013e318167ab1f. PMID 18349191
- [Background] Zimmermann M, Feibicke T, Keyl C, Prasser C, Moritz S, Graf BM, Wiesenack C. Accuracy of stroke volume variation compared with pleth variability index to predict fluid responsiveness in mechanically ventilated patients undergoing major surgery. Eur J Anaesthesiol. 2010 Jun;27(6):555-61. doi: 10.1097/EJA.0b013e328335fbd1. PMID 20035228
- [Background] Forget P, Lois F, de Kock M. Goal-directed fluid management based on the pulse oximeter-derived pleth variability index reduces lactate levels and improves fluid management. Anesth Analg. 2010 Oct;111(4):910-4. doi: 10.1213/ANE.0b013e3181eb624f. Epub 2010 Aug 12. PMID 20705785
- [Background] Desebbe O, Boucau C, Farhat F, Bastien O, Lehot JJ, Cannesson M. The ability of pleth variability index to predict the hemodynamic effects of positive end-expiratory pressure in mechanically ventilated patients under general anesthesia. Anesth Analg. 2010 Mar 1;110(3):792-8. doi: 10.1213/ANE.0b013e3181cd6d06. PMID 20185658